CLINICAL TRIAL: NCT04033263
Title: Maintaining Oral Health With Bio-products: a Randomized, Cross-over, in Situ Study
Brief Title: Maintaining Oral Health With Bio-products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SNSF-Project-1904
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries; Dental Erosion
MeSH Terms: conditions — Dental Caries; Tooth Erosion | interventions — Water; Fluorides

STUDY DESIGN:
Intervention Model Description: Cross-over study, where all participants will use all treatments. The treatment order will be set at random.
Who Masked: Participant, Care Provider
Masking Description: Mouth rinses will be placed in coded bottles, and the investigator and patients will not know to which group they belong. This is a cross-over study, where all 12 participants will use all 4 rinses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo mouth rinse (Placebo Comparator): Placebo: Deionized water (serving as negative control)
  Interventions: Other: Mouth rinse 1
- Elmex mouth rinse (Active Comparator): Commercial mouth rinse used as gold standard in erosion studies: elmex® Erosion Protection solution (which contains 800 ppm Sn2+, as SnCl2, and 500 ppm F-, as NaF and AmF)
  Interventions: Other: Mouth rinse 2
- Plant extract A with fluoride (Experimental): Plant Extract A + Fluoride
  Interventions: Other: Mouth rinse 4
- Fluoride (Active Comparator): NaF Fluoride Rinse
  Interventions: Other: Mouth rinse 3

INTERVENTIONS:
Other: Mouth rinse 1 — Participants will use 10mL of the respective mouth rinse, swish in the mouth for 30 seconds and spit it out. This will be made twice a day, for a total of 5 days.
  Other Names: Water
  Arms: Placebo mouth rinse
Other: Mouth rinse 2 — Participants will use 10mL of the respective mouth rinse, swish in the mouth for 30 seconds and spit it out. This will be made twice a day, for a total of 5 days.
  Other Names: Elmex Erosion Protection mouth rinse
  Arms: Elmex mouth rinse
Other: Mouth rinse 3 — Participants will use 10mL of the respective mouth rinse, swish in the mouth for 30 seconds and spit it out. This will be made twice a day, for a total of 5 days.
  Other Names: Fluoride mouth rinse
  Arms: Fluoride
Other: Mouth rinse 4 — Participants will use 10mL of the respective mouth rinse, swish in the mouth for 30 seconds and spit it out. This will be made twice a day, for a total of 5 days.
  Other Names: Plant extract A and fluoride
  Arms: Plant extract A with fluoride

SUMMARY:
This study will follow a randomised, double-blind, cross-over design. Participants will use mouth rinses containing plant extracts and/or fluoride, as well as a mouth rinse containing only water (placebo). They will use oral appliances containing sterilized enamel and dentine slabs, which will be later collected for analyses.

The cross-over design will allow participants to use all rinses, allowing for a comparison between the rinses within each individual.

DETAILED DESCRIPTION:
This study will be made in three in situ parts. Participants will wear an oral appliance containing sterilized enamel and dentine slabs. During this experimental phase, they will use the designated mouth rinse. After this period, the investigators will remove the enamel and dentine slabs, and will also collect salivary pellicle and any bacterial biofilm forming on the participant's teeth. Participants will also donate saliva for proteomic analysis (protein profile) to verify if there are any differences in proteins in saliva to proteins in the pellicle. Throughout the whole study, all participants will use standardized oral hygiene products.

The experimental mouth rinses contain plant extracts that could interact with salivary proteins and influence the salivary pellicle and oral biofilm, thus bringing positive results against tooth (enamel and dentine) demineralisation.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy young adults of both sexes, with normal salivary flow, with no cavitated caries lesions, no gingivitis or periodontal disease, no severe erosive tooth wear, and no other serious general or oral conditions.
* Participants will have signed an informed consent form.

Exclusion Criteria:

* Presenting oral diseases or conditions, such as untreated cavitated caries lesions, gingivitis or periodontitis, severe erosive tooth wear, etc.
* Participants who are under orthodontic treatment (wearing braces),
* Contraindications to the mouth rinses under study, e.g. known hypersensitivity or allergy to the investigational product,
* Participants using drugs that cause hyposalivation,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Individuals suffering from clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Specific exclusions for the disease under study,
* Specific concomitant therapy washout requirements prior to and/or during study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Enamel mineral loss | End of the study arm, expected to be after 1 week of using the mouth rinse
  Hardness of enamel slabs (Knoop hardness)
Dentine mineral loss | End of the study arm, expected to be after 1 week of using the mouth rinse
  Profilometry of dentine specimens (step height in µm)

SECONDARY OUTCOMES:
Identification of which proteins are present in the participants' saliva | End of the study arm, expected to be after 1 week of using the mouth rinse
  Proteomic analyses of the saliva (list of proteins present)
Identification of which proteins are present in the participants' salivary pellicle | End of the study arm, expected to be after 1 week of using the mouth rinse
  Proteomic analyses of the salivary pellicle (list of proteins present)
Thickness of the salivary pellicle | End of the study arm, expected to be after 1 week of using the mouth rinse
  Measured using TEM (mineralization measured in Delta Z)
pH of the participants' biofilm | End of the study arm in part 3, expected to be after 1 day of using the mouth rinse
  Measured in vivo after using the mouth rinses (pH)
Identification of the bacteria in the biofilm | End of the study arm in part 3, expected to be after 1 day of using the mouth rinse
  Measured after collecting the biofilm (list of bacterial species)
How many bacteria are adhered to the biofilm | End of the study arm in part 3, expected to be after 1 day of using the mouth rinse
  Measured after collecting the biofilm (bacteria quantity)

CONTACTS AND LOCATIONS:
Overall Officials: Thiago S Carvalho, PD Dr, Principal Investigator — University of Bern
Locations (1):
- Univesity of Bern (Klinik für Zahnerhaltung, Präventiv- und Kinderzahnmedizin), Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No